CLINICAL TRIAL: NCT01122355
Title: Comparison of Fenofibrate and Niacin in Patients With Hypertriglyceridemia and Low High-Density Lipoprotein (HDL)-Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sang Hak Lee/associate professor, Yonsei University, College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0530
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Hypertriglyceridemia With Low HDL-cholesterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- niacin arm (Active Comparator)
  Interventions: Drug: lipid modification
- fenofibrate arm (Active Comparator)
  Interventions: Drug: lipid modification

INTERVENTIONS:
Drug: lipid modification — 1) fenofibrate 160 mg po for 16 weeks, 2) niacin 500 mg po for 4 weeks, niacin 1000 mg po for 4 weeks, niacin 1500 mg po for 8 weeks

SUMMARY:
The purpose of the study is to compare the efficacy and tolerability of fenofibrate 160 mg and niacin 1500 mg in patients with hypertriglyceridemia and low HDL-cholesterol. The primary end point is the percent change of apoB/A1 and the secondary end points are other lipid parameters and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Triglyceride 150-500 mg/dL and HDL-cholesterol < 45 mg/dL after 8 week dietary run in period
* 20-79 years old

Exclusion Criteria:

* Low-density lipoprotein (LDL)-cholesterol ≥ 130 mg/dL without any lipid-modifying drug
* History of cerebrovascular or cardiovascular diseases
* Creatinine > 2.0 mg/dL
* Transaminase > 2x upper limit of normal
* Gall bladder disease
* Cancer
* Pregnant or breast feeding women
* History of adverse events associated with test drugs

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
percent change of apoB/A1 | after 16 weeks of drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hak Lee, Principal Investigator — professor of division of Cardiology